CLINICAL TRIAL: NCT05778188
Title: A Phase 2, Two-Stage, Randomized, Double-Blind, Placebo-Controlled, Multiple-Ascending Dose Study to Evaluate the Safety, Tolerability, Pharmacokinetics, and Preliminary Efficacy of RLS-0071 in Newborns With Moderate or Severe Hypoxic-Ischemic Encephalopathy Undergoing Therapeutic Hypothermia With Long-Term Follow-Up
Brief Title: A Study to Evaluate the Safety, Tolerability, Pharmacokinetics, and Preliminary Efficacy of RLS-0071 in Newborns With Moderate or Severe Hypoxic-Ischemic Encephalopathy Undergoing Therapeutic Hypothermia
Acronym: STAR
Status: Recruiting | Phase: Phase 2 | Type: Interventional
Sponsor: ReAlta Life Sciences, Inc. (Industry)
Collaborators: Premier Research (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: RLS-0071-202
Record Dates: First submitted 2023-03-03; First posted 2023-03-21 (Actual); Last update posted 2025-10-24 (Actual); Status verified 2025-10

CONDITIONS: Hypoxic-Ischemic Encephalopathy
Keywords: Birth Asphyxia; Anoxic brain injury
MeSH Terms: conditions — Hypoxia-Ischemia, Brain; Asphyxia Neonatorum | interventions — RLS-0071

STUDY DESIGN:
Intervention Model Description: Two-Stage, Randomized, Double-Blind, Placebo-Controlled, Multiple-Ascending Dose Study
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Masking Description: The blinded study team members (eg, Investigators and study staff) and participants' parent(s)/legal guardian(s) will be blinded to treatment group assignments throughout the study.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (2):
- RLS-0071 (Experimental): Doses of RLS-0071 to be administered every 8 hours (q8h), for a total of 10 doses over 72 hours.
  Interventions: Drug: RLS-0071
- Placebo (Placebo Comparator): Doses of sterile saline (sodium chloride, 0.9%) to be administered every 8 hours (q8h), for a total of 10 doses over 72 hours.
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: RLS-0071 — RLS-0071 (unit strength 10 mg/mL) will be administered by infusion for a dose level of 3 or 10 mg/kg. Planned infusion duration is 10 minutes for all dose levels.
  Arms: RLS-0071
Drug: Placebo — Placebo control (commercial sterile saline) will be administered by infusion at a volume matched to RLS-0071 (3 or 10 mg/kg). Planned infusion duration is 10 minutes for all matched dose levels.
  Arms: Placebo

SUMMARY:
Hypoxic-ischemic encephalopathy (HIE) affects approximately 4,000 to 12,000 persons annually in the United States. Mortality from HIE has been reported up to 60%, with at least 25% of survivors left with significant neurocognitive disability. Despite this vital unmet medical need, no pharmacological adjunct or alternative therapy has proven beneficial in improving outcomes in neonatal HIE.

RLS-0071 is a novel peptide being developed for the treatment of neonatal HIE. This study is designed to evaluate the safety and tolerability of RLS-0071 in the treatment of newborns with moderate or severe HIE.

DETAILED DESCRIPTION:
This is a Phase 2, two-stage, multisite, randomized, double-blind, placebo-controlled, multiple-ascending dose study of RLS-0071 to assess the safety, tolerability, pharmacokinetics (PK), and preliminary efficacy in newborns with moderate or severe HIE undergoing therapeutic hypothermia.

In Stage 1, participants will receive either ascending doses of RLS-0071 or a matched volume of placebo for 72 hours in addition to standard of care treatment, including therapeutic hypothermia. During and after the dosing period, participants will be monitored and assessed for safety evaluations through Day 14. After completion of Stage 1, participants will transition to Stage 2 of the study for long-term observation until participants reach 24 months of age.

The first cohort subsets, consisting of Cohort 1a (moderate HIE) and 1b (severe HIE), will receive a dose of 3 mg/kg RLS-0071 or a matched volume of placebo every 8 hours (q8h). A Data Safety Monitoring Board (DSMB) will review available clinical safety and PK data from Cohort 1 subsets with completed study intervention, and make a recommendation on whether to escalate the dose for moderate and severe HIE cohorts. The Sponsor will consider the DSMB recommendation to make their decision on dose escalation in addition to their own evaluation of all available safety and PK data. If the decision is made to escalate, Cohort 2 subsets (2a [moderate] and 2b [severe]) will be recruited to receive an escalated dose of RLS-0071 (10 mg/kg) or a matched volume of placebo. Following the completion of study intervention for each Cohort 2 subset (2a [moderate] or 2b [severe]), the DSMB will review available safety and PK data and make a recommendation whether to expand enrollment for Cohort 2+ (2a+ [moderate] or 2b+ [severe]) at 10 mg/kg RLS-0071 or a matched volume of placebo.

ELIGIBILITY:
Inclusion Criteria:

1. ≥ 36 weeks gestation.
2. Sentinel event prior to delivery such as abruption, tight nuchal cord, uterine rupture, profound bradycardia, shoulder dystocia, or cord prolapse or other acute event likely attributable for newborn depression at delivery or an acute change in the fetal status with a clinical presentation consistent with an acute sentinel event with no clearly defined etiology.
3. Moderate or severe encephalopathy based on at least one risk of encephalopathy criterion (a) and one clinical signs of encephalopathy criterion (b):

   1. Risk of encephalopathy (either):

      * Blood gas drawn within 1 hour of birth, either arterial blood gas (ABG) or venous blood gas (VBG) (cord or infant) with pH ≤ 7.0 OR base deficit ≥ 16 mmol/L.

      OR
      * appearance, pulse, grimace, activity, and respiration (APGAR) score ≤ 5 at 10 minutes OR
      * The infant required assisted ventilation ≥ 10 minutes after birth (ie, endotracheal, mask ventilation, or continuous positive airway pressure [CPAP]).
   2. Clinical signs of encephalopathy (either/both):

      * Moderate/Severe encephalopathy on National Institute of Child Health and Human Development assessment.
      * Evidence of seizures (clinical and/or electroencephalogram).
4. Be eligible to receive therapeutic hypothermia.
5. Active whole-body cooling to be started prior to 6 hours of age (passive cooling is permitted prior to active whole body cooling).
6. Product of a singleton pregnancy.
7. Written informed consent obtained from parent or legal guardian.

Exclusion Criteria:

1. Inability to enroll in the study and initiate the first dose of RLS-0071 within 10 hours of life.
2. Known major congenital and/or chromosomal abnormality(ies).
3. Severe growth restriction (birth weight ≤ 1800 g).
4. Prenatal diagnosis of brain abnormality or hydrocephalus.
5. Patient's head circumference is < 30 cm.
6. 10-minute APGAR score < 2, if available.
7. Infants suspected of overwhelming sepsis or congenital infection based on the Investigator's clinical consideration at the time of enrollment.
8. Persistent severe hypotension unresponsive to inotropic support (requiring >2 inotropes, not inclusive of hydrocortisone).
9. Persistent severe hypoxia in the setting of 100% fraction of inspired oxygen (FiO₂) and unresponsive to nitric oxide or requiring extracorporeal membrane oxygenation (ECMO).
10. Severe disseminated intravascular coagulation with clinical bleeding.
11. Neonatal encephalopathy believed to be due to a cause other than perinatal hypoxia (ie, other than HIE).
12. Moribund infants for whom withdrawal of care being considered.
13. Suspected or confirmed fetal alcohol syndrome or suspected substance withdraw seizures.
14. Any other condition that the investigator may consider would make the patient ineligible for the study or place the patient at an unacceptable risk (Note: this criterion would include a clinically significant [eg, Grade 3 or 4] intracranial hemorrhage).

Max Age: 10 Hours | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 42 (Estimated)
Dates: Start 2023-07-27 (Actual); Primary Completion 2026-04 (Estimated); Study Completion 2026-04 (Estimated)

PRIMARY OUTCOMES:
Frequency and severity of adverse events (AEs) and serious adverse events (SAEs) by treatment group at Day 14 | Day 1 to Day 14
  Number of participants with AEs and SAEs graded between Grade 1 (mild in severity) and Grade 5 (death related to AE).
Frequency and severity of events of special interest and SAEs by treatment group at 24 months | Day 1 to 24 months
  Number of participants with events of special interest and SAEs graded between Grade 1 (mild in severity) and Grade 5 (death related to AE).
  Events of special interest are: autoimmune disorder, persistent hypotension, persistent pulmonary hypertension, acute kidney injury, major venous thrombosis, severe intracranial hemorrhage, pulmonary hemorrhage, culture proven sepsis, necrotizing enterocolitis, severe thrombocytopenia, hepatic dysfunction, hyperbilirubinemia, coagulopathy, hypocalcemia, cerebral palsy, developmental or speech delay, learning disability, and visual or hearing impairment.
Frequency of premature discontinuation by treatment group due to AEs at Day 14 | Day 1 to Day 14
  Number of participants who prematurely discontinue from the study due to AEs
Acute brain injury at Day 4, assessed through magnetic resonance imaging (MRI), using a standardized scoring system | Day 4
  Brain injury MRI score includes scoring extent of injury across 4 domains (Grey matter, White matter/cortex, Cerebellum, and Additional). A score of 0 indicates a normal brain MRI, whereas the maximum score of 57 indicates extensive bilateral injury.
Acute brain injury at Day 12, assessed through magnetic resonance imaging (MRI), using a standardized scoring system | Day 12
  Brain injury MRI score includes scoring extent of injury across 4 domains (Grey matter, White matter/cortex, Cerebellum, and Additional). A score of 0 indicates a normal brain MRI, whereas the maximum score of 57 indicates extensive bilateral injury.

SECONDARY OUTCOMES:
Composite of mortality and neurodevelopmental impairment (NDI) at 24 months | Day 1 to 24 months
Mortality at 3, 6, 12, 18, and 24 months | Day 1 to 3, 6, 12, 18, and 24 months
  Number of participants alive at each timepoint
Number of participants with clinically significant laboratory abnormalities, events of special interest, and SAEs at 3, 6, 12, and 18 months | Day 1 to 3, 6, 12, and 18 months
Neurocognitive developmental outcome assessed by Bayley-4 at 24 months of age | 24 months
  The Bayley Scales of Infant and Toddler Development (4th Edition) consists of 5 subdomains: the Cognitive, Language, Motor, Social-Emotional, and Adaptive Behavior scales. Cognitive, Language, and Motor domains include a total of 264 items, each ranked between 0-2 (where 0 is not present and 2 is mastery); the Social-Emotional and Adaptive Behavior domains are assessed through caregiver questionnaires.
Neurodevelopmental growth impact: Diagnosis of cerebral palsy at 24 months of age | 24 months
  Number of participants diagnosed with cerebral palsy
Neurodevelopmental growth impact: Grading of cerebral palsy by using the Gross Motor Function Classification System-Expanded and Revised (GMFCS-E&R) at 24 months of age | 24 months
  The GMFCS is a 5-level classification system for children and young people with cerebral palsy, where Level 1 indicates ability to walk without limitations and Level 5 indicates reliance on a manual wheelchair.
Number of participants diagnosed with mild, moderate, or severe visual impairment and hearing impairment | Day 1 to 24 months
Number of days of supplemental nutritional support required | Day 1 to 24 months
Seizure occurrence | Day 1 to Day 14
  Discrete number of seizures recorded
Total seizure burden (total number of minutes seizing as measured by continuous electroencephalogram [EEG]) during hospitalization | Day 1 to Day 14
Electrical activity abnormality scoring as measured by EEG | Day 1 to Day 14
Impact on infant and family wellness, assessed by the Mother-to-Infant Bonding Scale (MIBS) | 3 and 12 months
  The MIBS is a 9-item questionnaire, with total scores ranging from 0 to 27. A high score indicates weaker mother-to-infant bonding.
Impact on infant and family wellness, assessed by the Parenting Stress Index, 4th Edition Short Form (PSI-4-SF) | 3, 12, and 24 months
  The PSI-4 is a 36-item questionnaire focusing on three domains: Parental Distress, Parent-Child Dysfunctional Interaction, and Difficult Child, which combine to form a Total Stress scale. Scores are assessed following conversion into percentile ranks. Scores falling in the 90th or higher percentile indicate clinically significant parenting stress.
Quality of life assessment over the first 24 months of life | Day 4 to 24 months
  A quality of life questionnaire will be used to collect information regarding the care of the aging child over the first 24 months of life.

OTHER OUTCOMES:
PK parameters of RLS-0071 at multiple-ascending doses: Cmax | Day 1 to Day 5
  Maximum serum concentration observed (Cmax) of RLS-0071
PK parameters of RLS-0071 at multiple-ascending doses: Ctrough | Day 1 to Day 5
  Concentration observed prior to subsequent or final dosing (Ctrough) of RLS-0071
PK parameters of RLS-0071 at multiple-ascending doses: Area under the curve | Day 1 to Day 5
  Area under the curve (AUC) of RLS-0071 concentration in serum
Number of participants diagnosed with epilepsy during the first 2 years of life | Day 1 to 24 months
Number of participants requiring anti-seizure medications during the first 2 years of life | Day 1 to 24 months
Brain injury MRI score at Day 4 and Day 12 for the white matter injury domain | Day 4 and Day 12
  Brain injury MRI score white matter domain includes the following items scored: cortex, cerebral white matter, optic radiations, corpus callosum, punctate white matter lesions, and parenchymal hemorrhage. The maximum white matter subscore is 21, indicating extensive bilateral injury.
Brain injury MRI score at Day 4 and Day 12 for the grey matter injury domain | Day 4 and Day 12
  Brain injury MRI score grey matter domain includes the following items scored: thalamus, basal ganglia, posterior limb of the internal capsule, brainstem, perirolandic cortex, and hippocampus. The maximum white matter subscore is 23, indicating extensive bilateral injury.
Number of days of mechanical ventilatory support required | Day 1 to Day 14 (or until discharge from hospital, if later)
  Duration until ability to breathe without assistance
Number of participants with pulmonary hypertension | Day 1 to 24 months
Number of days spent in the Neonatal Intensive Care Unit and number of days spent in the hospital | Day 1 to Day 14 (or until discharge from hospital, if later)
Severity of organ reperfusion injury as measured by clinical laboratory assessments: liver enzymes | Day 1 to Day 14
Severity of organ reperfusion injury as measured by clinical laboratory assessments: serum creatinine | Day 1 to Day 14
Severity of organ reperfusion injury as measured by synthetic liver function | Day 1 to Day 14

CONTACTS AND LOCATIONS:
Locations (15):
- United States (15):
  - Study Site 016, Little Rock, Arkansas
  - Study Site 013, Orange, California
  - Study Site 020, San Diego, California
  - Study Site 019, San Diego, California
  - Study Site 001, Gainesville, Florida
  - Study Site 018, Miami, Florida
  - Study Site 010, Orlando, Florida
  - Study Site 014, Indianapolis, Indiana
  - Study Site 012, Lexington, Kentucky
  - Study Site 002, Boston, Massachusetts
  - Study Site 006, St Louis, Missouri
  - Study Site 003, Durham, North Carolina
  - Study Site 021, Cleveland, Ohio
  - Study Site 022, Fort Worth, Texas
  - Study Site 005, Morgantown, West Virginia

IPD SHARING:
Plan to Share IPD: No